CLINICAL TRIAL: NCT02256891
Title: Arthroscopic Rotator Cuff Repair Using Standard Double Row Technique With Platelet Rich Fibrin Membrane vs. Standard Double Row Technique: A Randomized Blinded Outcomes Study
Brief Title: Rotator Cuff Repair Using Standard Double Row Technique With Platelet Rich Fibrin Membrane vs. Standard Double Row Technique
Acronym: RCRPRFM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 04100-11-C
Record Dates: First submitted 2014-08-04; First posted 2014-10-06 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2015-10

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff tear; Rotator cuff injury; Shoulder pain; Shoulder injury
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Shoulder Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double Row (Experimental): Double Row
  Interventions: Procedure: Double Row
- Double Row with PRFM (Experimental): Double Row with PRFM
  Interventions: Device: PRFM; Procedure: Double Row

INTERVENTIONS:
Device: PRFM
  Arms: Double Row with PRFM
Procedure: Double Row

SUMMARY:
This study is a single-blind, randomized study evaluating the 6 month and 2 year outcomes of patients treated with arthroscopic rotator cuff repair using one of two techniques. One technique used is the standard double row repairs utilizing medial and laterally based anchor fixation and the other technique is the standard double row repairs utilizing medial and laterally based anchor fixation with the use of plateley rich fibrin membrane (PRFM). It is hypothesized that patients undergoing the surgery with the PRFM will report a higher quality of life than the patients that do not receive this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a rotator cuff tear as determined by clinical examination and diagnostic imaging (MRI)
* Patient undergoes arthroscopic rotator cuff repair
* Age 18 or older

Exclusion Criteria:

Pre-operative exclusion criteria

* Patient has had a previous arthroscopic rotator cut repair
* A previous diagnosis of Rheumatoid Arthritis
* Evidence of major joint trauma, infection, avascular necrosis, chronic dislocation, inflammatory or degenerative glenohumeral arthropathy, frozen shoulder, or previous surgery of the affected shoulder,
* Evidence of significant rotator cuff arthropathy with superior humeral translation and acromial erosion diagnosed by x-ray or other investigations,
* Medical device that would exclude the patient from having a MRI, including a pacemaker, cardiac defibrillator, aneurysm clips, carotid artery clamp, neurostimulator, insulin or infusion pump, implanted drug infusion device, bone growth/fusion stimulator, or ear implant.
* Major medical illness (life expectancy less then 2 years or unacceptably high operative risk),
* Inability to speak or read English
* Psychiatric illness that precludes informed consent.
* Pregnant patients.
* Age 17 or younger
* Unwillingness to be followed for 2 years.
* Bilateral Rotator cuff tear confirmed by clinical exam and MRI
* Patients enrolled in the study who demonstrate retear on clinical exam and MRI, then elect for a repeat surgery.

Intra-operative exclusion criteria (Note: This information will be collected during the chart audit and patients will be excluded from the study at that time.)

* Irreparable cuff tears or tears extending into the subscapularis or teres minor
* Isolated teres minor or subscapularis tears.
* Inelastic and immobile tendon which cannot be advanced to articular margin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TRIA Orthopaedic Center, Bloomington, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Double Row With PRFM: Double Row with PRFM
  PRFM
  Double Row
Period: Overall Study
Arm/Group | Double Row | Double Row With PRFM
Started | 55 | 42
Completed | 43 | 29
Not Completed | 12 | 13
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 7 | 3
Not completed — Screen Fail | 5 | 4
Not completed — Equipment Malfunction | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Double Row Only: Double Row
- Double Row With PRFM: PRFM
- Total: Total of all reporting groups
Arm/Group | Double Row Only | Double Row With PRFM | Total
Number analyzed (Participants) | 55 | 42 | 97
Age, Continuous [Mean (Full Range); unit: years] | 53.00 [34 to 73] | 58.64 [42 to 75] | 56.15 [34 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 15 | 39
  Male | 31 | 27 | 58
Region of Enrollment [Number; unit: participants]
  United States | 55 | 42 | 97

OUTCOME MEASURES:

1. Primary Outcome: Return to Function
Description: The Western Ontario Rotator Cuff Index total score is on a scale of 0-2100; where 0 is the best score and 2100 is the score. There is a discrepancy between overall number of participants analyzed for this measure when compared to the participant flow module. More patients completed a baseline measure than those that completed the entire study.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 44 | 32
units on a scale | 1257.45 (396.07) | 1106.31 (393.78)

2. Primary Outcome: Return to Function
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 40 | 31
units on a scale | 371.38 (312.18) | 297.13 (221.21)

3. Primary Outcome: Return to Function
Description: Western Ontario Rotator Cuff Index
Time Frame: 24 months
Population: The Western Ontario Rotator Cuff Index total score is on a scale of 0-2100; where 0 is the best score and 2100 is the score. There is a discrepancy between overall number of participants analyzed for this measure when compared to the participant flow module. More patients completed a 24 month measure than those that completed the entire study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 41 | 28
units on a scale | 174.8 (254.41) | 103.11 (144.03)

4. Other Pre Specified Outcome: Spraspinatus Strength Measurements
Description: Strength of supraspinatus in newton meters with a hand held dynomometer. Three trials were recorded and an average taken. Data is reported as measured by % of uninvolved. Average of strength measures for involved/average of strength measures for uninvolved x 100.
Time Frame: Baseline
Population: There is a discrepancy between overall number of participants analyzed for this measure when compared to the participant flow module. More patients completed a baseline measure than those that completed the entire study.
Measure: Mean (Standard Deviation); unit: percentage of uninvolved
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 44 | 32
percentage of uninvolved | 45.4 (34.2) | 51.8 (32.3)

5. Other Pre Specified Outcome: MRI
Description: MRI was used to determine size of the defect in the proximal to distal, humeral to bursal, superior to inferior direction in all four tendons. All post operative rotator cuffs were described using the MRI rating system of Sugaya. This classification distinguishes 5 outcomes of rotator cuff repair based on integrity of the tendon determine by post operative MRI. Type I demonstrates the repaired rotator cuff has sufficient thickness and homogeneously low intensity on each image; Type II sufficient thickness with a partial high intensity area; Type III insufficient thickness without discontinuity, Type IV the presence of a minor discontinuity in more than one slice of each image suggestive of small tear; Type V the presence of a major discontinuity on each image suggestive of a large tear.
  Higher grades are worse radiographic outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 42 | 27
scores on a scale | 3.21 (1.07) | 2.74 (1.02)

6. Other Pre Specified Outcome: Supraspinatus Strength Measurements
Description: as for outcome 4
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of uninvolved
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 40 | 27
percentage of uninvolved | 73.0 (29.0) | 81.0 (26.0)

7. Other Pre Specified Outcome: Supraspinatus Strength Measurements
Description: as for outcome 4
Time Frame: 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of uninvolved
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 40 | 28
percentage of uninvolved | 101.0 (53.0) | 96.0 (17.0)

8. Other Pre Specified Outcome: Infraspinatus Strength Measurements
Description: Strength of infraspinatus in newton meters with a hand held dynomometer. Three trials were recorded and an average taken. Data is reported as measured by % of uninvolved. Average of strength measures for involved/average of strength measures for uninvolved x 100.
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of uninvolved
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 44 | 32
percentage of uninvolved | 73.6 (67.4) | 73.7 (24.3)

9. Other Pre Specified Outcome: Infraspinatus Strength Measurements
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of uninvolved
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 40 | 27
percentage of uninvolved | 90.0 (33.0) | 96.0 (22.0)

10. Other Pre Specified Outcome: Infraspinatus Strength Measurements
Description: as for outcome 8
Time Frame: 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of uninvolved
Arm/Group | Double Row | Double Row With PRFM
Number analyzed (Participants) | 40 | 28
percentage of uninvolved | 102.0 (23.0) | 104.0 (13.0)

ADVERSE EVENTS:
Time Frame: 24 month
Description: 24 month visit
Arm/Group | Double Row | Double Row With PRFM
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/42
Other Adverse Events (participants affected / at risk) | 9/55 | 2/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Row (N=55) | Double Row With PRFM (N=42)
Oncological (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Cancer
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Optomological (Eye disorders) | 1 (1) | 0 (0)
ENT (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Dermatological (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0)
Neurological (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A disadvantage is the majority of the tears are small or medium sized. These have a higher intrinsic healing and as such may not require platelet augmentation to afford a successful outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No